CLINICAL TRIAL: NCT06658366
Title: In Vivo Accuracy of Digital Intraoral Scans/Optical Impression Systems for the Production of Full-Arch Impressions
Brief Title: The Accuracy of Intraoral Scanning Systems for Full-Arch Impressions Is Examined in 10 Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-00618
Record Dates: First submitted 2024-07-25; First posted 2024-10-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-06

CONDITIONS: Full-arch Impression
Keywords: accuracy; intra oral scan; full-arch impression; conventional and optical impression of the teeth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Comparison conventional impression vs. digital impression (Other): The investigators would like to investigate the accuracy of various intraoral scanning systems. For this a conventional impression is taken from all patients to generate a reference model, which is then compared to full-arch impressions from various digital intraoral scanning systems.
  The examination is carried out in the same way for all participants.
  Interventions: Diagnostic Test: impression of the teeth

INTERVENTIONS:
Diagnostic Test: impression of the teeth — Only conventional and digital impressions (comparable with taking videography) are taken of the patients teeth.

SUMMARY:
For several decades now, modern procedures have allowed dentists to capture your teeth using digital cameras. This digital procedure is increasingly replacing traditional impressions with a viscous mass that hardens in the mouth.

In the following study, the investigators want to find out whether the accuracy of these modern methods is comparable to the classic impression technique.

Three conventional impressions are taken for this purpose, and multiple digital impressions are also taken with each of the intraoral scanners. The impressions are then compared with each other. This allows the accuracy of the different intraoral scanners to be determined.

DETAILED DESCRIPTION:
In summary, this study intends to address the need for comprehensive in vivo research on the accuracy of intraoral impression methods, especially in the context of modern digital technologies. By comparing various digital and conventional methods, this research will offer valuable information to guide dental practitioners in choosing the most precise and reliable techniques for their clinical applications.

The following study design is planned:

The study is non-randomised. The study setup is monocentric. At the beginning of the session, 3 conventional impression each of the upper and lower jaw is taken. After 8 hours the impression is moulded by a dental technician with a SuperHard plaster (type 4).After 48 hours of setting time the plaster-model is scanned with a lab scanner (inEos X5, Dentsply Sirona) to generate a .stl-file that is comparable to the following digital impressions.

This is followed by 6 digital impressions of the upper and lower jaw and the associated bite registration in habitual occlusion, divided between two experienced practitioners (3 upper, 3 lower jaw scans, 3 bite registrations per practitioner) with the 8 different intra oral scanners. In total, 6 conventional (3 upper, 3 lower jaw impressions), 48 digital impressions and 48 bite registration are taken. If it is not possible to take all the impressions in one session, a new conventional impression is taken at the start of each new session, so that a daily updated reference model is always available. Minimizing bias is achieved, by using the intra oral scanners according to the manufacturers instructions.

The number of scans was calculated as part of a power analysis based on previous study results and should therefore be meaningful.

The selection of scanners represents a heterogeneous selection of devices currently on the market. The scanners come from different price categories and use different optical measuring principles.

The precision measurement is carried out by comparing the impressions within and between the tested groups (precision and trueness respectively). For that, the scans will be exported to STL & PLY format (depending on the scanning device) and imported into evaluation programs (Dentexion, Dentexion and Control X, Geomagic). The evaluation process follows the ISO 5725-1 criteria. After superimposition of the mesh surfaces according to the best-fit alignment, the distances will be measured point-to-point using the signed nearest neighbor method and sorted into a histogram. From that, the distance measure for each pairwise surface superimposition will be calculated from the (90%-10%)/2 percentile value.

ELIGIBILITY:
Inclusion Criteria:

* All genders, minimum age for participation is 18 years
* Good general health and healthy dental conditions (gaps with a maximum of 1 missing tooth are permitted)
* Written consent after informed consent discussion is available

Exclusion Criteria:

* participants under the age of 18
* Addicts or participants with impaired cognitive abilities that do not allow the participant to assess the scope of the study
* participants suffering from periodontitis (pathological tooth mobility could falsify the study results)
* Maximal mouth opening less than 3.5 cm
* participants who wear large reconstructive works and/or have a free-end situation from at least the 2nd premolar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Accuracy measurement of digital impressions performed with optical impression systems are primary endpoints | It is intended that all impressions take place within half a day, the accuracy measurement should be carried out within 6 weeks.
  The accuracy of the intraoral scanners (primary endpoint) is analyzed on the basis of precision and trueness. The unit of measure used is the same (μm).
  The trueness of each test group is assessed by superimposing each scan with the reference model data set. The precision is calculated as the mean difference between all superimpositions within one test group.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Center for Dental Medicine, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
The ethics application, which has already been approved, contains clear provisions on data protection. There is no provision for data to be passed on; accordingly, the investigators must protect all personal data and may not pass it on to third parties.

REFERENCES:
- [Result] Ender A, Attin T, Mehl A. In vivo precision of conventional and digital methods of obtaining complete-arch dental impressions. J Prosthet Dent. 2016 Mar;115(3):313-20. doi: 10.1016/j.prosdent.2015.09.011. Epub 2015 Nov 6. PMID 26548890